CLINICAL TRIAL: NCT00637442
Title: Continuous Arterial Spin Labeling (CASL) MRI for Monitoring and Prediction of Drug Therapy in Alzheimers Disease (AD)
Acronym: CASL-AD-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Bonn (Other)
Collaborators: Federal Ministry of Health, Germany (Other Government)
Responsible Party: Frank Jessen, MD, University Hospital, Bonn
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: University Bonn
Record Dates: First submitted 2008-02-15; First posted 2008-03-18 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CASL-MRI (Experimental): Drug monitoring with CASL-MRI for new diagnosed patients with mild to moderate Alzheimer's Disease treated with Reminyl
  Interventions: Drug: Reminyl retard

INTERVENTIONS:
Drug: Reminyl retard — retard tablets once a day WEEK1-4: 8mg; WEEK 5-8: 16mg, WEEK 9-24: 24mg

SUMMARY:
Examination of the correlation between the cerebral bloodflow and the clinical change under treatment with Reminyl retard® and the prediction of clinical change by measuring the cerebral bloodflow in patients with mild to moderate Alzheimer's Disease

ELIGIBILITY:
Inclusion Criteria:

* Possible Alzheimer's Disease according to ICD-10 and NINCDS-ADRDA
* Underwritten study consent
* No treatment with acetylcholinesterase inhibitors
* Mini-Mental-State Examination: 12-25 points
* Age: 50-80 Years
* Orale contraception for women of child-bearing age

Exclusion Criteria:

* Mental Disorders
* Other Diseases of the CNS
* Severe Illness
* Contraindication for MRI-Scan
* Contraindication for Galantamin (Reminyl retard®)
* Participation at other clinical trials

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Cerebral perfusion | baseline and after 12 weeks

SECONDARY OUTCOMES:
Change of Alzheimer Disease Assessment Scale, cognitive part (ADAScog) | baseline, after 12 and 24 weeks
Alzheimer's Disease Functional Assessment and Change Scale (ADFACS) | baseline, after 12 and 24 weeks
Neuropsychiatric Inventory (NPI) | baseline, after 12 and 24 weeks
Mini-Mental-Status-Examination (MMSE) | baseline, after 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frank Jessen, MD, Principal Investigator — University Bonn
Locations (1):
- Department of Psychiatry, University Bonn, Bonn, Germany